CLINICAL TRIAL: NCT03745066
Title: A Post-Market Registry of the BioFreedomTM Biolimus A9TM Coated Coronary Stent System
Brief Title: BioFreedom French Registry
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Biosensors Europe SA (Industry)
Collaborators: European Cardiovascular Research Center (Network)
Responsible Party: Sponsor
Other Study IDs: 18-EU-01
Record Dates: First submitted 2018-11-05; First posted 2018-11-19 (Actual); Last update posted 2021-04-26 (Actual); Status verified 2021-04

CONDITIONS: Coronary Artery Disease
Keywords: coronary artery disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Prospective, observational multi-center registry to be conducted at up to 25 French interventional cardiology centers. Patients will be eligible once they have received at least one BioFreedomTM DCS as per standard clinical practice and will be followed for up to 2 years post PCI for data collection.

The purpose of the registry is to explore the safety and effectiveness of the BioFreedomTM DCS in standard clinical practice in France and to serve as part of Post Market Surveillance.

DETAILED DESCRIPTION:
Prospective, observational multi-center registry to be conducted at up to 25 French interventional cardiology centers. Patients will be eligible once they have received at least one BioFreedomTM DCS as per standard clinical practice and will be followed for up to 2 years post PCI for data collection.

The registry will be purely observational and will not interfere with physician's decisions relating to stent selection or indication for treatment.

The purpose of the registry is to explore the safety and effectiveness of the BioFreedomTM DCS in standard clinical practice in France and to serve as part of Post Market Surveillance.

ELIGIBILITY:
Inclusion Criteria:

* Patients treated with one or more BioFreedom™ DCS .Patients who agree to comply with the follow up requirements. .Patients with a life expectancy of > 1 year at time of consent. .Patients eligible to receive dual anti platelet therapy (DAPT).
* Patients who have signed an Informed Consent

Exclusion Criteria:

* Patients unable or unwilling to give documented informed consent
* Patients taking part in another interventional trial which has not completed follow-up for the primary endpoint .Patient has received an additional stent different from a BioFreedom™ DCS stent during the index procedure.
* Pregnant or breastfeeding women
* Planned surgery within 6 months of percutaneous coronary intervention (PCI) unless dual antiplatelet therapy is maintained throughout the peri surgical period for non HBR patients
* Planned surgery within 1 month of percutaneous coronary intervention (PCI) unless dual antiplatelet therapy is maintained throughout the peri surgical period for HBR patients
* Patients under judicial protection, tutorship or curatorship

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This observational registry is open to all patients with coronary artery disease treated by percutaneous coronary intervention (PCI) with one or more BioFreedom™ DCS within the indications of the Instructions for Use.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2019-04-04 (Actual); Primary Completion 2021-04-30 (Estimated); Study Completion 2022-04-27 (Estimated)

PRIMARY OUTCOMES:
DOCE | 1 year
  Device-oriented composite endpoint (DOCE) at 12 months defined as composite of cardiovascular death (CD), myocardial infarction (MI) not clearly attributable to a non-target vessel and clinically driven target lesion revascularization (cd-TLR).

SECONDARY OUTCOMES:
All-cause mortality | 12-month and 24-month
  1. All-cause mortality, CD, non-cardiovascular and undetermined death in hospital and at 12 and 24 months
Patient-oriented composite endpoint (POCE) at 12 and 24 months | 12 months and 2 years
  Patient-oriented composite endpoint (POCE) at 12 and 24 months defined as all-cause mortality, any stroke, any MI (including nontarget vessel territory) and any revascularization.
Composite of Cardiovascular Death (CD) at 12 and 24 months | 12 months and 2 years
  Composite of CD, MI and definite/probable stent thrombosis (ST) at 12 and 24 months.
Definite/probable ST at 12 and 24 months | 12 months and 24 months
  Definite/probable ST at 12 and 24 months
Target Vessel Failure defined at 12 and 24 months | 12 months and 24 months
  Target Vessel Failure (TVF) defined as CD, target-vessel-related MI, and Target vessel revascularization (TVR) at 12 and 24 months
Target Lesion Failure at 12 and 24 months | 12 months and 24 months
  Target Lesion Failure (TLF) defined as CD, target-vessel-related MI, and clinically driven TLR at 12 and 24 months
Clinically driven TLR at any follow-up time point | Inclusion, 12 months and 24 months
  Clinically driven TLR at any follow-up time point
Clinically driven TVR at any follow-up time point | Inclusion, 12 months and 24 months
  Clinically driven TVR at any follow-up time point
Any revascularization | within 24 months following the index procedure
  Any revascularization within 24 months following the index procedure, unless they are planned within the 1st month
Stroke, disabling and non-disabling. | Inclusion, 12 months and 24 months
  Stroke, disabling and non-disabling.
BARC 3 to 5 bleeding | Inclusion, 12 months and 24 months
  BARC 3 to 5 bleeding

CONTACTS AND LOCATIONS:
Overall Officials: Janusz Lipiecki, MD, Principal Investigator — Clinique des Dômes; Philippe Garot, MD, Principal Investigator — ICPS, Massy
Locations (6):
- France (6):
  - Clinique Des Dômes, Clermont-Ferrand, Cedex 2
  - at Hôpital Privé Claude Galien ICPS, Quincy-sous-Sénart, Essonne
  - Clinique de Fontaine, Fontaine-lès-Dijon
  - Centre Hospitalier General, Haguenau
  - Clinique Saint Martin, Pessac
  - CHU Toulouse Rangeuil, Toulouse